CLINICAL TRIAL: NCT02775838
Title: Measurements of Kidney Perfusion After Transplantation by Intraoperative Fluorescence Angiography
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Collaborators: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Ulrich Rother, Dr. med. Ulrich Rother, University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPY-Kidney
Record Dates: First submitted 2016-04-13; First posted 2016-05-18 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Indocyanine Green

ARMS (1):
- kidney transplantation (Experimental): Intravenous injection of Indocyanine Green in patients receiving kidney transplantation
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — perioperative application of Indocyanine green (ICG)

SUMMARY:
Aim of this clinical study is to establish a novel technique, the so called intraoperative fluorescence angiography, for kidney graft perfusion visualization during the transplant procedure.

DETAILED DESCRIPTION:
Additional to the common transplant procedure, measurements of the graft perfusion should be established in two ways. Firstly, each kidney should be measured by a common duplex ultrasound measurement to assess the resistance index (RI) in the three poles of the kidney (upper, middle, lower pole). Secondly, intraoperative fluorescence angiography is going to be performed. Therefore, the camera of the fluorescence angiography system (SPY Elite System, Novadaq, USA) is positioned over the organ, and the fluorescence dye (ICG) is applicated intravenously. The aim will be to correlate the fluorescence angiography findings with the RIs and therefore to establish valuable fluorescence parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving kidney transplantation
* Deceased donor and living donor transplantations

Exclusion Criteria:

* Allergy against indocyanine green
* Iodine allergy
* Contrast allergy
* Penicillin allergy
* Allergic diathesis
* Liver insufficiency
* Pregnancy
* Hyperthyreosis
* Pulmonary arterial hypertension

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation of intraoperative SPY Perfusion Parameters with short-term outcome of the graft function | 24 Months
  The intraoperative fluorescence parameters (Ingress, Ingressrate, Egress, Egressrate) will be correlated with the creatinine level of the first 10 postoperative days.

SECONDARY OUTCOMES:
Evaluation of the ideal ICG dosage for intraoperative kidney perfusion | 6 Months
Correlation of intraoperative measured resistance indices with fluorescence parameters (Ingress, Ingressrate, Egress, Egressrate) | 12 Months
Correlation of graft rejection episodes and fluorescence parameters | 24 Months
Correlation of fluorescence parameters with numbers of dialysis needed during the first 10 postoperative days | 24 Months

OTHER OUTCOMES:
Correlation of intraoperative fluorescence parameters of the ureter with ureter anastomosis complications postoperatively | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Rother, Dr. med., Principal Investigator — University of Erlangen, Vascular Surgery; Kai Nowak, Prof. Dr. med., Principal Investigator — University of Mannheim, General Surgery
Locations (2):
- Germany (2):
  - University of Erlangen, Vascular Surgery, Erlangen
  - University of Mannheim, General Surgery, Mannheim

REFERENCES:
- [Derived] Gerken ALH, Nowak K, Meyer A, Weiss C, Kruger B, Nawroth N, Karampinis I, Heller K, Apel H, Reissfelder C, Schwenke K, Keese M, Lang W, Rother U. Quantitative Assessment of Intraoperative Laser Fluorescence Angiography With Indocyanine Green Predicts Early Graft Function After Kidney Transplantation. Ann Surg. 2022 Aug 1;276(2):391-397. doi: 10.1097/SLA.0000000000004529. Epub 2020 Dec 30. PMID 33394595